CLINICAL TRIAL: NCT06210152
Title: Influence of Radial Extracorporeal Shockwave Therapy on Achilles Tendon on Ankle Functionality
Brief Title: Does Radial Extracorporeal Shockwave Therapy Applied to the Achilles Tendon Influence Ankle Functionality?
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hyunjoong Kim (Other)
Responsible Party: Sponsor-Investigator, Hyunjoong Kim, Investigator, Sahmyook University
Organization: Sahmyook University (Other)
Other Study IDs: 2-1040781-A-N-012021092HR
Record Dates: First submitted 2023-12-20; First posted 2024-01-18 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Radial Extracorporeal Shockwave Therapy
  Interventions: Device: Radial Extracorporeal Shockwave Therapy
- Sham Extracorporeal Shockwave Therapy
  Interventions: Device: Sham Extracorporeal Shockwave Therapy

INTERVENTIONS:
Device: Radial Extracorporeal Shockwave Therapy — Radial Extracorporeal Shockwave Therapy (rESWT) was administered using the Masterpuls® MP200 device (Storz Medical AG, Tägerwilen, Switzerland). Participants were seated with their calves exposed. A coupling gel was applied to the Achilles tendon area and, adhering to the 90° application rule, a 15-mm applicator was used in both transverse and diagonal patterns at the myotendinous junction, extending across the muscle belly using a smoothing motion. Each session involved the delivery of 1000 pulses at a frequency of 10Hz and an air pressure setting of 1.0 bar.
  Groups: Radial Extracorporeal Shockwave Therapy
Device: Sham Extracorporeal Shockwave Therapy — Sham Extracorporeal Shockwave Therapy (rESWT) was administered using the Masterpuls® MP200 device (Storz Medical AG, Tägerwilen, Switzerland). Participants were seated with their calves exposed. A coupling gel was applied to the Achilles tendon area and, adhering to the 90° application rule, a 15-mm applicator was used in both transverse and diagonal patterns at the myotendinous junction, extending across the muscle belly using a smoothing motion. In each session, the device was held against the achilles tendon without being powered on.
  Groups: Sham Extracorporeal Shockwave Therapy

SUMMARY:
Radial Extracorporeal Shockwave Therapy has been shown to restore shortened muscles and normalize fibrotic tissues in muscles or fascia. Shockwave therapy can soften fibrotic tissues and alleviate pain. While there are various methods to relax muscles and fascia, radial extracorporeal shockwave therapy can achieve good results in a short treatment time. Although there is research on the pain-related effects of radial extracorporeal shockwave therapy for conditions such as plantar fasciitis and knee osteoarthritis, there is a lack of literature on its functional effects. Therefore, this study aims to investigate the improvement of ankle functionality through the application of radial extracorporeal shockwave therapy.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who have ankle-related pain scores of 0 to 2 on the Numeric Pain Rating Scale (NPRS).
* Individuals with no functional impairment in the ankle.

Exclusion Criteria:

* Individuals who have undergone surgical procedures such as ankle joint arthrodesis.
* Individuals showing signs of functional impairment in ankle functionality.
* Individuals with ankle-related pain rated above 3 on the NPRS.
* Individuals with acute ankle fractures.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The recruitment of participants for the study is planned to take place in Han-nam-dong and at Sahmyook University in Seoul, Republic of Korea. Potential participants selected through recruitment documents will be enrolled upon meeting the eligibility criteria. After providing a comprehensive explanation of the study, those who voluntarily agree to participate will be recruited.
Sampling Method: Probability Sample
Enrollment: 33 (Estimated)
Dates: Start 2024-01-10 (Estimated); Primary Completion 2024-01-17 (Estimated); Study Completion 2024-01-19 (Estimated)

PRIMARY OUTCOMES:
Jump height | Immediate change from baseline after intervention
  The Single-Leg Vertical Jump is measured using the OptoGait System (Microgate, S.R.L, Bolzano, Italy, 2010) to determine maximum height, flight time, and ground contact time. Higher jumps, longer flight times, and shorter ground contact times indicate improved single-leg vertical jump performance. The setup involves placing two parallel bars embedded with sensors on either side and positioning a camera in front. Participants, with their shoes removed, enter between the bars. They are instructed to "Please jump as high as you can, five times," with the command given loudly. After five jumps, the collected data are processed using the OptoGait software (Version 1.5.0.0, Microgate, S.R.L). Jump height (cm) is calculated from the maximum jump height in OptoGait.
flying time | Immediate change from baseline after intervention
  The Single-Leg Vertical Jump is measured using the OptoGait System (Microgate, S.R.L, Bolzano, Italy, 2010) to determine maximum height, flight time, and ground contact time. Higher jumps, longer flight times, and shorter ground contact times indicate improved single-leg vertical jump performance. The setup involves placing two parallel bars embedded with sensors on either side and positioning a camera in front. Participants, with their shoes removed, enter between the bars. They are instructed to "Please jump as high as you can, five times," with the command given loudly. After five jumps, the collected data are processed using the OptoGait software (Version 1.5.0.0, Microgate, S.R.L). Flying time (msec) is calculated as hover time when jumping in OptoGait.
contact time | Immediate change from baseline after intervention
  The Single-Leg Vertical Jump is measured using the OptoGait System (Microgate, S.R.L, Bolzano, Italy, 2010) to determine maximum height, flight time, and ground contact time. Higher jumps, longer flight times, and shorter ground contact times indicate improved single-leg vertical jump performance. The setup involves placing two parallel bars embedded with sensors on either side and positioning a camera in front. Participants, with their shoes removed, enter between the bars. They are instructed to "Please jump as high as you can, five times," with the command given loudly. After five jumps, the collected data are processed using the OptoGait software (Version 1.5.0.0, Microgate, S.R.L). Contact time (msec) is calculated by OptoGait as the time on the floor before jumping.

CONTACTS AND LOCATIONS:
Locations (1):
- Sahmyook University, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes